CLINICAL TRIAL: NCT05106244
Title: The Application of Remote Real-Time Guidance System in Home Care of Patients With PICC or PORT
Brief Title: Remote Real-Time Guidance System in Home Care of Patients With PICC or PORT
Acronym: RRTGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-300
Record Dates: First submitted 2021-09-16; First posted 2021-11-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-09

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- family self-nursing mode (Experimental)
  Interventions: Other: Real-Time Guidance of Home Care for Patients with PICC or PORT
- hospital nursing mode (No Intervention)

INTERVENTIONS:
Other: Real-Time Guidance of Home Care for Patients with PICC or PORT — the experimental group adopted the family self-nursing mode, mainly by the patients' family members to observe the catheter and do regular nursing, and the specialist nurses provided remote real-time online guidance to monitor the family nursing of central venous catheter. The procedures are as follows: (1) make nursing videos recorded by central venous catheter specialist nurses; (2) evaluate the nursing operation ability of the patients' family members and carry out relevant training and health education, repeat until they are qualified; (3) distribute nursing guidance prescriptions and maintenance manuals for central venous catheters; (4) provide online simulated realistic nursing video materials; (5) provide real-time telephone audio and video connection to complete remote nursing guidance. (6) set up a home nursing volunteer service group, establish a doctor-patient exchange group by using Wechat and other media.
  Arms: family self-nursing mode

SUMMARY:
Clinical treatment of digestive tract tumor patients often need chemotherapy before and after operation, most chemotherapy drugs will cause harm to patients, prone to leakage, leading to tissue necrosis. The construction of deep venous channels can protect the blood vessels of patients and reduce their pain. PICC and PORT have become a new clinical treatment technology, and have become the mainstream mode of long-term intravenous indwelling. Although the central venous catheterization technology has many advantages, it also has some limitations. Because of its long-term existence, periodic nursing needs to be carried out, such as correct flushing, sealing, replacement of film and so on. Incorrect care or failure to come to the hospital on time may lead to abnormal use of the catheter or shortening of service life, resulting in some unexpected pain. Under the influence of COVID-19 's epidemic situation, it becomes more difficult and unrealistic for patients to come to hospital regularly for nursing. During the epidemic, patients need more safe and effective care at home. In order to help patients with good central venous catheter nursing at home, this study intends to apply remote professional real-time guidance technology to home nursing care of PICC and PORT tumor patients. Through on-site practical operation training, video explanation materials of long-distance on-line decomposition steps and real-time telephone audio connection guidance are provided to enable patients' families to quickly learn to master nursing techniques, so as to achieve safe and effective self-care at home.

DETAILED DESCRIPTION:
From January 2022 to October 2022, 200 patients with digestive tract tumors with indwelling PICC or PORT in the inpatient department of oncology surgery in First Affiliated Hospital of Xian Jiaotong University were randomly divided into control group (hospital nursing mode) and experimental group (family self-nursing mode) . The specific methods were as follows: 2-1 the control group adopted regular nursing mode after catheterization. The patients were mainly given on-site catheterization nursing by specialist nurses, and health consultation and guidance were carried out during the period of catheterization. 2-2 the experimental group adopted the family self-nursing mode, mainly by the patients' family members to observe the catheter and do regular nursing, and the specialist nurses provided remote real-time online guidance to monitor the family nursing of central venous catheter. The specific operation procedures are as follows: (1) make nursing videos recorded and reviewed by central venous catheter specialist nurses (video production is carried out separately for different central venous access devices from different manufacturers, as well as follow-up training steps). (2) evaluate the nursing operation ability of the patients' family members and carry out relevant training and health education, including hand washing, aseptic concept, matters needing attention in removing the film, flushing and sealing techniques, and local observation points at the puncture point, etc., repeatedly strengthen the training of key links and conduct assessment until the participants are qualified; (3) distribute nursing guidance prescriptions and maintenance manuals for central venous catheters. (4) provide online simulated realistic nursing video materials, nursing video materials are decomposed in detailed steps, each step is equipped with detailed language explanation and explanation, and the key links are reminders or warnings. It is convenient for patients' families to learn and master quickly; (5) provide real-time telephone audio and video connection to complete remote nursing guidance. (6) set up a home nursing volunteer service group, which is composed of nursing team members led by central venous catheter specialist nurses, establish a doctor-patient exchange group by using Wechat and other media, and provide nursing outpatient information of each central venous catheter in the area. Improve family nursing failure remedial measures, provide necessary guidance and help, and timely feedback. The normal service life of the catheter, the infection rate of the catheter puncture point, the catheter occlusion rate, the nursing experience and satisfaction of the patients and their families were compared between the two groups. Statistical processing: the data were analyzed by SPSS22.0 software. The measurement data are expressed as mean ± standard deviation, t-test is used, counting data is expressed as rate (%), and 2 test or Fisher exact probability method is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastric cancer or colorectal cancer with indwelling central venous catheter (PICC or PORT)
* Age ≥18 years and ≤75 years
* Normal cognitive function
* Be informed of and actively cooperate with this study

Exclusion Criteria:

* Suffering from psychological disorders and not able to communicate normally
* Unable to cooperate due to other factors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Average level of service life of the catheter | up to 10 months
  Average length of service life of PICC or PORT
Incidence of puncture point infection | up to 10 months
  Incidence of puncture point infection of PICC or PORT
Incidence of catheter occlusion | up to 10 months
  Incidence of catheter occlusion of PICC or PORT
Degree of satisfaction of patients and their families | up to 10 months
  a satisfaction survey of patients and their families, using a self-designed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhang, Doctor, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China